CLINICAL TRIAL: NCT00363779
Title: Microarray Analysis of the Effect of Cyclosporine Therapy on Gene Expression Patterns in Large Granular Lymphocytic Leukemia
Brief Title: Effect of Cyclosporine Therapy on Gene Expression in Patients With Large Granular Lymphocyte Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to low accrual and the investigator left the NIH.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thomas Waldmann, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060177; 06-C-0177
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-06

CONDITIONS: Large Granular Lymphocytic Leukemia; LGL Leukemia
Keywords: Large Granular Lymphocyte (LGL); LGL; Leukemia; Cyclosporine; Microarray; Gene Expression; Cyclosporin; Large Granular Lymphocyte Leukemia; LGL Leukemia
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic; Leukemia | interventions — Cyclosporine; Gene Expression Profiling; Microarray Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LGL Patients administered cyclosporine (Experimental): Large Granular Lymphocyte Leukemia (LGL) is a low grade non-Hodgkins lymphoma characterized by tissue invasion of the marrow, spleen, and liver. Cyclosporine 5-10 mg/kg/day was administered as an oral preparation given every 12 hours. Doses are adjusted to maintain a therapeutic level between 200-400 ng/ml.
  Interventions: Drug: Cyclosporine; Genetic: Gene expression analysis; Genetic: Microarray analysis; Other: Laboratory biomarker analysis

INTERVENTIONS:
Drug: Cyclosporine — An oral preparation given every 12 hours, 5-10 mg/kg/day in divided doses. Doses are adjusted to maintain a therapeutic level between 200-400 ng/ml. Levels will be checked twice weekly and once the patient has achieved steady state levels they shall be monitored once every 2 weeks. These therapeutic levels shall be maintained for 3 months.
  Other Names: Ciclosporin
Genetic: Gene expression analysis — A permutation test will be performed to examine whether the overall expression profile changes due to treatment. This will be done by comparing the number of significant genes to the distribution of this number if in fact there is no difference between pre-treatment and post-treatment gene expression.
Genetic: Microarray analysis — Gene expression profiling will be carried out on Affymetrix microarrays to compare pretreatment and posttreatment samples.
Other: Laboratory biomarker analysis — Analysis of differential gene expression profiles in patients with LGL leukemia treated with cyclosporine.

SUMMARY:
Background:

* Large granular lymphocyte (LGL) leukemia is a low-grade non-Hodgkin's lymphoma.
* LGL is associated with low numbers of white blood cells (leading to recurring infections), red blood cells (causing anemia) and platelets (causing abnormal bleeding).
* Cyclosporine (CSA) is an immunosuppressive drug that improves low blood cell counts in about 50 percent of patients with LGL leukemia.

Objectives:

* To identify what factors determine why cyclosporine works in some patients and not in others.
* To identify what causes low blood counts in LGL leukemia.

Eligibility: Patients 18 years of age and older with LGL leukemia.

Design:

* Patients have a medical history, physical examination blood tests, bone marrow biopsy and x-ray studies, including chest x-rays and computed tomography (CT) scans of the chest, abdomen and pelvis. Patients with an easily accessible enlarged lymph node have a node biopsy (removal of a small piece of tissue for microscopic examination).
* Patients take cyclosporine twice a day by mouth. Blood samples are taken at least weekly to adjust the cyclosporine dosing to maintain therapeutic serum levels.
* Patients undergo apheresis (collection of white blood cells) at a number of different time points in the study (maximum 6 times) to look at the differences in the leukemia cells before and during treatment with cyclosporine. For apheresis, blood is withdrawn through a needle in an arm vein and directed through a catheter (plastic tube) into a machine that separates it into its components. The white cells are extracted and the rest of the blood is returned through the same needle or through a second needle in the other arm.

DETAILED DESCRIPTION:
Background:

* LGL leukemia is a low grade non-Hodgkins Lymphoma characterized by tissue invasion of the marrow, spleen and liver
* Recurrent infections due to chronic neutropenia and transfusion-dependent anemia are the principal causes for initiation of therapy
* Approximately 50% of patients treated with cyclosporine (CSA) respond to treatment. CSA appears to correct the associated cytopenia without decreasing LGL numbers, suggesting it may inhibit LGL secretion of yet unidentified mediators of neutropenia and anemia.
* Analysis of differential gene expression profiles in patients with LGL leukemia treated with cyclosporine has the potential to detect as yet unidentified, therapeutic targets and possibly provide predictors of CSA responsiveness.

Objective:

* Identify changes in gene expression patterns induced by cyclosporine therapy in patients with LGL leukemia
* Identify differences between responding and non-responding patients

Eligibility:

-Patients with Large Granular Lymphocyte leukemia

Design:

* Patients will be treated with cyclosporine at a dose of 5-10mg/kg/day in divided doses, with doses adjusted to maintain a therapeutic serum level between 200-400ng/ml. These therapeutic levels shall be maintained for 3 months.
* Tumor response will be evaluated after 3 months therapy, the dose of CsA may then be tapered to that required to sustain a response or discontinued if no evidence of response, or after relapse.
* Blood sampling or Lymphapheresis for collection of circulating malignant cells will be performed at a number of different time points. Gene expression profiling will be carried out on Affymetrix microarrays to compare pretreatment and post-treatment samples.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. All patients must have a histologic or cytologic diagnosis of T-cell LGL leukemia as determined by the Laboratory of Pathology or Hematology at the Clinical Center, National Institutes of Health
  2. All patients must have hemocytopenias such as granulocyte count less than 1,200/ul, platelet count less than 100,000/ul or hemoglobin less than 10 g/dl, or require hematopoietic support (transfusion or colony stimulating factors) to maintain counts at these or higher levels.
  3. Patients must have measurable or evaluable disease
  4. Patients must have a creatinine of less than 2.0 mg/dl.
  5. Omission of cytotoxic chemotherapy for 3 weeks prior to entry into the trial is required. However, patients receiving stable corticosteroids will be eligible.
  6. Age greater than 18 years
  7. Karnofsky performance greater than 70%
  8. Patients must have a life expectancy of greater than 3 months.
  9. Patients must be able to understand and sign an Informed Consent form.
  10. All female patients must use adequate contraception during participation in this trial and for three months after completing therapy.

EXCLUSION CRITERIA:

1. Patients with uncontrolled hypertension
2. Pregnant and nursing patients are not eligible for the study as CSA crosses the placenta. Based on clinical use, premature births and low birth weight were consistently observed. Breast-feeding is contraindicated because CSA enters the blood milk and may possibly be administered to the child.
3. Underlying immunodeficiency state including human immunodeficiency virus (HIV) seropositivity.
4. Positive for antibodies to hepatitis C or positive for hepatitis B surface antigen,
5. Patients with serious intercurrent illnesses, concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious or metabolic disease of such severity that it would preclude the patients' ability to tolerate cyclosporine.
6. Patients who received cyclosporine for LGL leukemia previously and failed to respond.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Waldmann, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lamy T, Loughran TP Jr. Clinical features of large granular lymphocyte leukemia. Semin Hematol. 2003 Jul;40(3):185-95. doi: 10.1016/s0037-1963(03)00133-1. PMID 12876667
- [Background] Vie H, Chevalier S, Garand R, Moisan JP, Praloran V, Devilder MC, Moreau JF, Soulillou JP. Clonal expansion of lymphocytes bearing the gamma delta T-cell receptor in a patient with large granular lymphocyte disorder. Blood. 1989 Jul;74(1):285-90. PMID 2546620
- [Background] Lamy T, Dauriac C, Le Prise PY. Long-term survival in chronic granulocytic leukaemia. Br J Haematol. 1989 Oct;73(2):279. doi: 10.1111/j.1365-2141.1989.tb00270.x. No abstract available. PMID 2818949
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: US FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LGL Patients Administered Cyclosporine
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LGL Patients Administered Cyclosporine
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gene Expression Patterns
Description: The goal was to examine which genes had a 2-fold gene expression between pre-treatment (baseline) and post treatment (12 weeks). Genes significant at the 0.001 level will be considered as differentially expressed due to treatment.
Time Frame: Baseline and 12 weeks
Population: This outcome measure was not performed because there were insufficient data points to provide any statistical power.
Arm/Group | LGL Patients Administered Cyclosporine
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 3 months
Measure: Number; unit: Participants
Arm/Group | LGL Patients Administered Cyclosporine
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 3 yrs, 10 months
Arm/Group | LGL Patients Administered Cyclosporine
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGL Patients Administered Cyclosporine (N=5)
Infection with normal ANC or Grade 1 or 2 neutrophils-Lung (pneumonia) (Infections and infestations) | 1 (1)
Second malignancy-possibly related to cancer treatment (Specify) new abdominal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGL Patients Administered Cyclosporine (N=5)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 (2)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (7)
Alkaline phosphatase (Investigations) | 2 (3)
Bicarbonate, serum-low (Investigations) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 5 (10)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (2)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 1 (2)
Creatinine (Investigations) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (8)
Hemoglobin (Blood and lymphatic system disorders) | 3 (11)
Hypertension (Vascular disorders) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (5)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (2)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 4 (5)
Pain::Muscle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Platelets (Investigations) | 3 (6)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (9)
Tremor (Nervous system disorders) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (2)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As there were only 5 patients treated, the primary endpoints of this protocol were not met and there is not enough data generated for statistical analysis. This protocol is being terminated due to low accrual and the investigator leaving the NIH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No